CLINICAL TRIAL: NCT02178137
Title: Effect of Interventions on Progression of Knee Osteoarthritis - a Comparison of Effect of Glucosamine/Chondroitin or Diacerin Vs Placebo: Measured by Clinical, Radiological and Biochemical Parameters
Brief Title: Effect of Interventions on the Progression of Knee Osteoarthritis
Acronym: KAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Principal Investigator, Mansoor Ali Khan, Professor, Orthoepedics, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIH-Ortho-001
Record Dates: First submitted 2014-06-27; First posted 2014-06-30 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Osteo Arthritis of the Knees
MeSH Terms: interventions — diacerein; Glucosamine; Chondroitin; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glucosamine/Chondroitin (Active Comparator): Glucosamine/Chondroitin twice a day for a daily total dose of 1500 mg of Glucosamine and 1200 mg of Chondroitin.
  Tablets will have 750 mg Glucosamine Sulphate and 600 mg of Chondroitin Sulphate. These will be taken twice a day after breakfast and dinner.
  Interventions: Drug: Glucosamine/Chondroitin
- Diacerien (Active Comparator): Diacerien 50 mg twice a day in capsule form. To be taken twice a day after breakfast and dinner
  Interventions: Drug: Diacerien
- Placebo pill (Placebo Comparator): Placebo tablets with Zinc sulfate twice a day. These will contain pharamacologically non active ingredients (Usually expedients).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diacerien
  Other Names: Artrodar; Dirtacetylrhein
  Arms: Diacerien
Drug: Glucosamine/Chondroitin
  Arms: Glucosamine/Chondroitin
Drug: Placebo
  Other Names: Zinc Sulphate
  Arms: Placebo pill

SUMMARY:
There has been intensive search for a substance that can have disease-modifying activity for osteoarthritis. A number of medications have been reported to be of benefit on slowing progression of knee OA. This trial will be the first head to head comparison of these medications.

Patients aged between age 40 to 65 will be enrolled. Patients will be assessed clinically using two scoring systems, the WOMAC index for knee arthritis and the SF 36 for overall physical and mental health. The knee X rays will be assessed on Kellgren and Lawrence grading and will also be measured for joint space narrowing at follow up. The response to arthritis medications on slowing down cartilage loss will be measured biochemically with COMP levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged between 40 to 65 years with mild to moderate osteoarthritis of the knees.
* Patients should have history of knee pain for at least 6 months and on the majority of days during the preceding month
* Each joint will be scored separately so one patient with bilateral knee osteoarthritis will be counted as 2 knees.
* The osteoarthritis will be graded on basis of clinical score as well as seen on appropriately positioned x rays using the Kellgren and Lawrence grading. (Tibio femoral osteophytes of at least 1 mm, Kellgren Lawrence grading of 2 or 3)
* Patients with diabetes are sent to the diabetes clinic and are included once their HbA1c level becomes normal.
* Patients giving Informed consent

Exclusion Criteria:

* Patients with severe end stage tricompartmental osteoarthritis of the knees .
* Presence of uncontrolled systemic disease like chronic liver and renal disease
* Patients with diagnosis other than osteoarthritis, such as knee arthritis due to rheumatoid disease, gout, post traumatic arthritis
* Patients with history of surgery to any knee will have that knee excluded
* Pregnant or lactating mothers
* Patients with chronic anaemia
* Patients who get an injection in their affected knee

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC score at 24 months in comparison to baseline score | baseline, 24 months
  Hypothesis:- At least one of the intervention drug will result in an improvement of at least 20 points on the WOMAC score at end of 2 years as compared to the placebo when compared to base line score
Change to the SF-36 score at 24 months in comparison to baseline score | 24 months
  Hypothesis: At least one of the intervention drugs will result in an improvement of at least 20 points at end of two years when assessed using the SF36 total score as compared to the standard therapy placebo when compared with baseline score
Mean differences in blood serum COMP levels of study arms | 24 months

SECONDARY OUTCOMES:
Change in WOMAC score at 6 months in comparison to baseline score | 6 months
Change in WOMAC score at 12 months in comparison to baseline score | 12 months
Change in WOMAC score at 18 months in comparison to baseline score | 18 months
Change to the SF-36 score at 6 months in comparison to baseline score | 6 months
Change to the SF-36 score at 12 months in comparison to baseline score | 12 months
Change to the SF-36 score at 18 months in comparison to baseline score | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor A Khan, MBBS, Principal Investigator — The Indus Hospital
Locations (1):
- The Indus Hospital, Karachi, Sindh, Pakistan